CLINICAL TRIAL: NCT02532218
Title: Randomized Evaluation of ARI-3037MO, to Suppress LDL Cholesterol in Patients With Dyslipidemia
Brief Title: Evaluation of ARI-3037MO, to Suppress LDL Cholesterol in Patients With Dyslipidemia
Acronym: REASCEND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arisaph Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI-3037MO-005
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2015-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): ARI-3037MO (niacin analog) 3g bid for 24 wks
  Interventions: Drug: ARI-3037MO
- Placebo (Placebo Comparator): Matching Placebo 3g bid for 24 wks
  Interventions: Drug: ARI-3037MO

INTERVENTIONS:
Drug: ARI-3037MO — Lipid lowering treatment Statins

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ARI-3037MO compared to placebo in reducing low-density lipoprotein cholesterol (LDL-C) levels in subjects with dyslipidemia.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized, double-blinded, controlled clinical trial. The study will compare two arms: ARI-3037MO 3 g BID vs. placebo.

Subjects who sign informed consent will be enrolled and will undergo all Visit 1 assessments. Following evaluation of Visit 1 laboratory assays, eligible subjects will receive a phone call (Visit 2) during which they will be instructed to begin the lifestyle modification and enter a 4- to 6-week lead-in period (6-week wash-out period for subjects to wash out of non-statin lipid-lowering therapy [subjects may remain on statins during this period], 4 weeks for subjects receiving statins only or not receiving any lipid-lowering therapy), followed by a qualifying fasting LDL-C measurement at Visit 3. After the lead-in period, if the LDL-C level at Visit 3 is not ≥ 100 mg/dL, an additional week will be allowed for another qualifying measurement at a subsequent visit (Visit 3.1). If performed, the LDL-C level at Visit 3.1 must be ≥ 100 mg/dL in order for the subject to continue participation in the study. Qualifying subjects will be randomized in a 1:1 manner at Visit 4 to one of two arms of the double-blind, 24-week efficacy and safety assessment phase. Randomization will be stratified by background statin therapy status at Visit 1 (yes/no). Baseline lipid levels will be defined as lipid levels at Visit 4. End-of-study lipid levels will be defined as the lipid levels at Visit 7 (Week 24).

A final closeout and safety assessment visit will be held at 26 weeks post randomization (Visit 8).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at screening.
2. Women of childbearing potential, must agree to use 2 medically accepted, effective methods of birth control. Females who are postmenopausal must have been postmenopausal for > 1 year if they wish not to use contraceptives. If postmenopausal status is questionable, the subject's follicle-stimulating hormone level must be elevated and consistent with postmenopausal levels (i.e., > 40 IU/L); otherwise these subjects must agree to use contraceptives listed above.
3. Male subjects with sexual partners of childbearing potential must be surgically sterile or using an acceptable method of contraception from the time of screening through 12 weeks after last dose of study drug to prevent pregnancy in a partner.
4. Female subjects of childbearing potential (including females with questionable postmenopausal status) must have a negative pregnancy test prior to dosing.
5. LDL-C level: ≥ 100 mg/dL.
6. Triglycerides (TG) ≤ 300 mg/dL.
7. High-density lipoprotein cholesterol (HDL-C) level < 45 mg/dL in men and < 50 mg/dL in women.
8. Subject understands the trial requirements and the treatment procedures, is willing to comply with all protocol-required follow-up evaluation and provides written informed consent
9. Subjects will be managed according to current standard of care. Subjects taking statin therapy will remain on their statin background therapy and must be on a stable dose, defined as no changes in the dose of statin in the 3 months prior to screening, and must be willing and able to remain on that dose for the duration of the study.

Exclusion Criteria:

1. Subjects treated with any statin at its maximally approved dose will be excluded from the study.
2. Body mass index (BMI) > 45 kg/m2.
3. Weight change ≥ 3 kg during the lead-in period.
4. Uncontrolled diabetes, defined as glycosylated hemoglobin (HbA1C) > 9.5%.
5. Contraindication to niacin treatment (prior flushing is not regarded as a contraindication to niacin treatment).
6. History of stroke, myocardial infarction, life-threatening arrhythmia, or having had coronary vascularization within 6 months before screening.
7. Thyroid-stimulating hormone ≥ 1.5 times the upper limit of normal (ULN).
8. Clinical evidence of hypothyroidism or thyroid hormonal therapy that has not been stable for ≥ 6 weeks before screening.
9. Creatine kinase concentration ≥ 3 times the ULN.
10. Known, active liver disease, including but not limited to

    1. Confirmed alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase ≥ 2 times the ULN, or bilirubin ≥ 1.5 times the ULN.
    2. Hepatitis C (anti-hepatitis C virus immunoglobulin G +).
    3. Hepatitis B (hepatitis B surface antigen +, anti-hepatitis B core antigen immunoglobulin M +).
11. Blood donation of ≥ 1 pint (0.5 L) within 30 days before screening or plasma donation within 7 days before screening.
12. Known nephrotic syndrome or ≥ 3 g/day proteinuria.
13. Past organ transplant or on a waiting list for an organ transplant.
14. Subject is currently receiving chemotherapy; or has received chemotherapy within the 30 days prior to screening; or is scheduled to receive chemotherapy during the course of the study.
15. Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 12 months.
16. Problems with substance abuse, which, in the opinion of the Investigator, might affect study compliance.
17. Planned procedure that may cause non-compliance with the protocol or confound data interpretation.
18. Participation in another investigational drug trial in the past 30 days or current participation in a device trial that has not reached its primary endpoint.
19. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study or within 12 weeks after last dose of study drug.
20. Estimated glomerular filtration rate < 60 mL/min/1.73 m2. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
LDL-c | 24 wks
  change in LDL cholesterol level

SECONDARY OUTCOMES:
HDL-c | 24 wks
  Change in HDL cholesterol
TG | 24 wks
  Change in triglyceride levels
HbA1C | 24 wks
  Change in hemoglobin A1C

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Catalina Reserch Institute, LLC, Chino, California
  - S&W Clinical Reserch, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonvile, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Sestron Clinical Research 833 Campbell Hill Street Suite 230, Marietta, Georgia
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Rochester clinical Research,Inc, Rochester, New York
  - Sterling Research Group Ltd, Cincinnati, Ohio
  - The Carl and Edyth Lindner Center for Reserch and education at the Christ Hospital, Cincinnati, Ohio
  - Metabolic and atherosclerosis Research center, Cincinnati, Ohio
  - IVA reserch, Cincinnati, Ohio
  - Sterling Research group, Ltd, Cincinnati, Ohio
  - Ohio Clinical Research-Lyndhurst, Lyndhurst, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - Willamette Valley Clinical studies, Eugene, Oregon
  - Health Research of Hampton Roads - Norfolk, Norfolk, Virginia
  - National Clinical Research inc, Richmond, Virginia
  - Raninier Clinical Reserach, Renton, Washington